CLINICAL TRIAL: NCT05767229
Title: Acute Hemodynamic Response to Carvedilol in Children With Clinically Significant Portal Hypertension.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-56
Record Dates: First submitted 2023-02-15; First posted 2023-03-14 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carvedilol for 1.5 hrs (Experimental): Carvedilol 0.2 mg/kg for 1.52 hrs
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Carvedilol 0.2 mg/kg for 1.5 hrs

SUMMARY:
Clinically significant portal hypertension (CSPH) is defined as Hepatic Venous Pressure gradient (HVPG) >10 mmHg. Patients with CSPH are at risk of developing esophageal varices and clinical decompensation (variceal bleeding, ascites, jaundice, encephalopathy), which mark the transition from compensated stage to a stage of the disease (decompensated) associated with higher mortality. HVPG is calculated by subtracting the free hepatic venous pressure (FHVP), a measure of systemic pressure, from the wedged hepatic venous pressure (WHVP), a measure of hepatic sinusoidal pressure. HVPG is surrogate marker in many clinical applications such as gold standard test to evaluate presence and severity of portal hypertension (PHT) diagnosis, risk stratification, monitoring of the patients on beta blockers. Non-selective beta-blockers like propranolol and carvedilol are indicated in adults for primary and secondary prophylaxis of variceal hemorrhage. Acute hemodynamic response to intravenous propranolol with HVPG values coming down to < 12 mm Hg or reduction to >20% from baseline have been shown to be associated with reduced long-term risk of variceal bleed. Portal Hypertension in biliary atresia (BA) occurs early and is due to recurrent cholangitis and portal sclerosis. HVPG in children is feasible and safe in children according to previous studies, however, there are no recommendations to suggest beta-blockers based on HVPG reduction in children. Hence, we are planning the current work to study the acute hemodynamic response to carvedilol in children with CSPH, and to compare the HVPG values in children with chronic liver disease.

DETAILED DESCRIPTION:
Aim: To study acute hemodynamic response Hepatic Venous Pressure Gradient (HVPG) reduction to <12 mm Hg or by ≥ 20% from initial value) to carvedilol in from 2 to 18 year of age children with Chronic liver disease.

Methodology Study population: All children (2-18) years of age with CLD as per inclusion and exclusion criteria

Study design: Prospective cohort

Baseline parameters that will be recorded:

* Baseline characteristics:
* History and etiology of liver disease
* Symptomatology, Evidence of decompensation (jaundice,organomegaly, encephalopathy, ascites, infections, variceal bleed etc)
* Clinical and demographic profile
* Variceal bleed, ascites, infections, hepatic encephalopathy, AKI
* Endoscopic findings:
* Esophageal varices
* Red colour signs
* Gastric varices
* Clinically significant varices
* Portal hypertensive gastropathy
* Liver and splenic stiffness
* Splenic Z-score - based on ultrasound measure of spleen (in cm) and calculation of Z-scores based on centiles from Indian children
* Anthropometric parameters:
* Weight for age
* Height for age
* Weight for length
* BMI
* Triceps skin fold thickness

Study period: 2 years

Sample size with justification: Since it is a pilot study we will take 40 patients

Methodology for HVPG measurement:

* 6-hour fasting
* procedure will be done either without sedation or minimal Sedation using propofol and ketamine
* Continuous ECG and Pulse-OX monitoring.
* 4 or 5 Fr venous introducer sheath will be places in right IJV using Seldinger technique under Doppler USG guidance
* Right or middle hepatic vein will be catheterized under fluoroscopic guidance with a 3 or 4 Fr Cobra angiographic catheter and a hydrophilic wire.
* The angiographic catheter will be exchanged with a 4 or 5 Fr occlusion balloon catheter
* All measurements will be recorded using a pressure transducer set linked to a multichannel recorder with a 50mmHg scale
* Zeroing: Before recording, the transducer will be placed at the level of right atrium (mid-axillary line) and kept it open to zero.
* FHVP will be measured by maintaining the tip of the catheter ''free'' in the hepatic vein, 1 to 3 cm from its opening into the IVC.
* WHVP will be measured while the catheter in hepatic vein and a balloon will be inflated at the tip of catheter. Adequate occlusion of the hepatic vein will be checked by slow injection of 2-5 mL of iodinated contrast (iodixanol iso-osmolar contrast medium, Visipaque 320 mgI/ml) with the catheter tip positioned in the mid/distal portion of the vein; typical ''wedged'' pattern, without reflux of the contrast or washout through communications with other hepatic veins will be considered confirmatory.
* Repeat testing will be done in children with HVPG >/= 10 mm Hg 90 minutes after giving carvedilol through nasogastric route.

Acute Hemodynamic response to oral carvedilol:

* Baseline heart rate and non-invasive BP monitoring (appropriate cuff).
* Following HVPG measurement, a single dose of carvedilol will be administered (0.2 mg/kg) via nasogastric route/oral and 90 minutes later, we will recheck heart rate, BP and HVPG. Percent change in HVPG will be calculated.
* Acute hemodynamic response is characterized as HVPG <12 mm Hg or reduction by >/=20%

Monitoring and Assessment:

1. All patients with esophageal varices or HVPG >10 mm Hg or both, will be started on oral Carvedilol 0.2 mg/kg/day, which will be increased every 3rd day upto 0.8 mg/kg/day to titre decrease in heart rate upto 25% from baseline.
2. Repeat UGIE after 6 months to see change in variceal status.

Statistical Analysis All the categorical variables will be expressed as frequencies, whereas continuous ones will be expressed as mean+ SD or median (IQR). Chi-square , Fisher's exact test and student's t-test will be applied for assessment of causality. Kaplan-Meier statistics will be done for survival and liver related morbidity besides this an appropriate analysis will be carried out at the time of data analysis like diagnostic test, logistic regression etc. Significance will be mentioned in the form of p-value <0.05.

Adverse effects:

* There are few side effects of beta blockers (carvedilol) like suppression of chronotropic effect, bronchospasm, hypoglycemia, exercise intolerance and hypotension and the patient will be carefully monitored for these for a duration of 6 hours post-procedure.
* Reversal of effect of carvedilol: In case of excessive bradycardia, hypotension or bronchospasm following measures will be taken:
* Bradycardia & hypotension: Intravenous atropine 1-2 mg +/- Intravenous glucagon 2.5-5 mg over 3-5 minutes, followed by continuous infusion at the rate of 1-5 mg/hour +/- Adrenaline / Dobutamine infusion as per weight adjusted dose.
* Bronchospasm: Nebulization with salbutamol/levosalbutamol/Adrenaline +/- intravenous aminophylline.

Stopping rule of study:

* Progression to exclusion criteria
* Adverse effects
* Potential liver transplant within 15 days

ELIGIBILITY:
Inclusion Criteria:

* All children 2-18 years of age with CLD defined as presence of either of the following histological evidence of advanced fibrosis more than F2 on METAVIR staging or radiological imaging suggestive (heterogeneous hepatic echotexture, irregular nodular liver and/or caudate hypertrophy). .
* Splenomegaly and/or platelets </= 100 (X10^3/mm3)
* Coming for upper gastrointestinal endoscopy for variceal screening
* Informed consent for HVPG and UGIE

Exclusion Criteria:

* Uncorrected heart defects (except small ASD)
* Cardiac conduction defects - arrythmias or heart block
* Interrupted inferior vena cava
* Situs inversus
* Patients who received beta-blockers in last 7 days
* Patients who received Octreotide infusion or bolus in last 7 days
* Variceal bleed in last 48 hours
* Shock or active sepsis
* Grade 2 /grade 3 ascites
* Severe hepatic impairment with MELD or PELD score >14
* Acute kidney injury (any grade)
* Hepatic encephalopathy (any grade)
* Known contraindications to propranolol in children:
* Hyper-reactive airway disease
* Hypertrophic cardiomyopathy
* Acute congestive heart failure

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Proportion of children with acute hemodynamic response 90 mins after carvedilol given through nasogastric route) in those with clinically significant portal hypertension. | 90 minutes
  Acute hemodynamic response (HVPG reduction to less than 12 mm Hg or by more than equals to 20% from initial value

SECONDARY OUTCOMES:
HVPG values in children (2-18 years age) with different etiologies of chronic liver disease. | Day 0
Proportion of children with presence of varices and clinically significant varices in children with HVPG more than equal to 10 in different etiologies of liver disease.. | Day 0
Proportion of children with presence of varices and clinically significant varices in children with HVPG less than 10 mm Hg in different etiologies of liver disease. | Day 0
Splenic Z-scores, Liver and splenic stiffness in children with HVPG more than equal to 10 or less than 10 mm Hg in different etiologies of liver disease. | Day 0
Bile acid levels in children with HVPG more than equal to 10 or less than 10 mm Hg in different etiologies of liver disease. | Day 0
Risk factors of acute hemodynamic response on univariate and multivariate binary logistic regression analysis. | Day 0
Change in the grading (low or high risk) of esophageal varices at 6 months after starting oral carvedilol in children with or without acute hemodynamic response. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided